CLINICAL TRIAL: NCT06880484
Title: Effect of Far-Infrared Emitting Socks on Neuropathic Pain, Nerve Conduction, and Quality of Life in Patients With Diabetic Peripheral Neuropathy: A Randomized Controlled Trial
Brief Title: Far-Infrared Socks for Neuropathic Pain and Nerve Function in Diabetic Patients
Acronym: FIR-DPN
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: TC Erciyes University (Other)
Responsible Party: Principal Investigator, Harun İN, Harun İn, MSc, Principal Investigator, TC Erciyes University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 1782/1762; 1782/1762 (Other: Erciyes Üniversitesi)
Record Dates: First submitted 2025-02-04; First posted 2025-03-17 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: Diabetic Peripheral Neuropathy (DPN)
Keywords: Diabetic Peripheral Neuropathy; Neuropathic Pain; Far-Infrared Therapy; Infrared Socks; Quality of Life; Diabetes Complications; Non-Pharmacological Treatment; Randomized Controlled Trial; Pain Management
MeSH Terms: conditions — Neuralgia; Diabetes Complications; Agnosia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental Group (Experimental): Patients will be selected from those attending endocrinology and neurology clinics or hospitalized and meeting the inclusion criteria. Participants will complete the Patient Information Form, LANSS Scale, and NePIQoL forms in a quiet room in the endocrinology ward. The Ankle Brachial Index will be evaluated to exclude peripheral arterial disease. If ENMG and lab findings are unavailable, patients will be referred for necessary tests. They will receive two pairs of FIR socks to be worn at least 8 hours daily, along with usage training. Contact information will be collected. Participants will be called three times to assess compliance and comfort via VAS. After three months, they will return for a final evaluation, including an ENMG scan by neurology specialists, and complete the LANSS Scale and NePIQoL forms again.
  Interventions: Device: Far-Infrared Radiation (FIR) Socks
- Placebo Socks Group (Placebo Comparator): Placebo group patients will be selected from those attending endocrinology and neurology clinics or hospitalized and meeting inclusion criteria. Participants will complete the Patient Information Form, LANSS Scale, and NePIQoL forms in a quiet room. The Ankle Brachial Index will be evaluated to exclude peripheral arterial disease. If ENMG and lab findings are unavailable, patients will be referred for necessary tests. They will receive two pairs of non-FIR socks to be worn at least 8 hours daily, along with usage training. Contact information will be collected. Participants will be called three times to assess compliance and comfort via VAS. After three months, they will return for a final evaluation, including an ENMG scan by neurology specialists, and complete the LANSS Scale and NePIQoL forms again.
  Interventions: Device: Placebo Socks

INTERVENTIONS:
Device: Far-Infrared Radiation (FIR) Socks — Participants in the experimental group will receive two pairs of Far-Infrared Radiation (FIR) emitting socks, designed to be worn for at least 8 hours per day over a 3-month period. These socks utilize FIR technology, which is hypothesized to improve circulation, reduce neuropathic pain, and enhance quality of life in patients with diabetic peripheral neuropathy (DPN). Participants will be educated on the proper use of the socks, provided with a usage protocol, and monitored for adherence via three follow-up phone calls assessing compliance and comfort using the Visual Analog Scale (VAS). At the end of the study, participants will undergo a follow-up Electroneuromyography (ENMG) evaluation, and pain and quality of life will be reassessed using the LANSS Scale and NePIQoL forms.
  Other Names: Far-Infrared Therapy Socks
  Arms: Experimental Group
Device: Placebo Socks — Participants in the placebo group will receive two pairs of non-FIR socks, which are visually identical to the FIR socks but lack FIR-emitting properties. They will follow the same 8-hour daily usage protocol for 3 months and receive the same education on sock usage. Compliance and comfort will be monitored through three follow-up phone calls, and assessments will be conducted using the VAS, LANSS Scale, and NePIQoL forms. At the end of the study, participants will undergo a final ENMG evaluation.This study aims to determine the effect of FIR socks on neuropathic pain, nerve conduction, and quality of life, using both subjective (pain scales) and objective (ENMG) measures.
  Other Names: Non-FIR Socks
  Arms: Placebo Socks Group

SUMMARY:
This study aims to evaluate the effectiveness of far-infrared radiation (FIR) emitting socks in improving neuropathic pain, nerve conduction, and quality of life in patients with diabetic peripheral neuropathy (DPN). It is the first comprehensive study in Turkey investigating FIR technology for DPN treatment and offers an alternative approach to traditional methods.The study will be conducted at Erciyes University Gevher Nesibe Hospital between February 2025 and June 2026 as a randomized controlled trial (RCT) with a triple-blind design. Participants will be assigned to either the FIR socks group or the placebo group, with both groups receiving two pairs of socks to wear daily. Assessments will include the Leeds Assessment of Neuropathic Symptoms and Signs (LANSS) Scale, the Neuropathic Pain Impact on Quality of Life (NePIQoL) questionnaire, and the Visual Analog Scale (VAS) for patient-reported outcomes. Electroneuromyography (ENMG) testing will also be performed before and after the intervention to assess nerve function.

This research is expected to provide clinical evidence on FIR socks as a non-pharmacological treatment for neuropathic pain, contributing to improved patient care and the development of innovative medical technologies in Turkey.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with diabetic peripheral neuropathy (DPN) with mild to moderate severity based on clinical evaluation.
* Oriented to person, place, and time (cognitively intact).
* Residing in Kayseri and receiving treatment in the city.
* HbA1C level below 8.5% during the study period.
* Non-smoker for at least 6 months.
* Not using neuropathic pain medication for at least 3 months before enrollment.
* Body Mass Index (BMI) between 25 - 35.
* Able to be contacted by phone for follow-up.
* Willing to participate and provide informed consent.

Exclusion Criteria:

* Presence of diabetic foot ulcers.
* Non-mobilized individuals (unable to walk independently).
* Severe peripheral artery disease (Ankle Brachial Index (ABI) < 0.4).
* Liver failure or renal failure (dialysis patients).
* Coronary artery disease.
* Candidates for surgery during the intervention period.
* Lower extremity arthroplasty or orthosis indication during the intervention period.
* Neurological or cognitive impairments (e.g., dementia, Alzheimer's disease).
* Receiving non-pharmacological treatment for diabetic peripheral neuropathy (DPN).
* Chronic alcohol or substance use.
* Severe anemia, vitamin B12 deficiency, or iron deficiency anemia.
* Recent changes in diabetes medication or newly diagnosed with diabetes.
* Neurological, cardiovascular, or orthopedic damage affecting the lower extremities.
* Use of cytotoxic or immunosuppressive agents or history of radiation therapy.
* Pregnant, breastfeeding, or attempting to conceive.
* Receiving physiotherapy at any point during the study period.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-02-02 (Actual); Primary Completion 2026-02-03 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Leeds Assessment of Neuropathic Symptoms and Signs (LANSS) Scale | The scale was filled in the baseline
  The Leeds Neuropathic Symptoms and Signs Assessment Scale (LANSS) was developed by Bennett (2001) and its Turkish validity and reliability study was conducted by Yücel et al. (2004). It is used clinically to differentiate neuropathic pain from nociceptive pain and consists of a five-item pain questionnaire (max: 16 points) and a two-item sensory assessment (max: 24 points). The pain questionnaire evaluates symptoms like tingling, paresthesia, skin color changes, electric shock sensations, and burning pain. The sensory section includes Allodynia and Pinprick tests; in the Allodynia test, a cotton wisp is applied to painful and non-painful areas-if discomfort is reported in the affected region, allodynia is considered present. If the total score is ≥12, pain is classified as neuropathic, while a score <12 indicates nociceptive pain. The scale has 82-91% sensitivity and 80-94% specificity when compared to clinical diagnosis.

SECONDARY OUTCOMES:
Neuropathic Pain Impact on Quality of Life (NePIQoL) | The scale was filled in the baseline
  The Neuropathic Pain Impact on Quality of Life Questionnaire (NePIQoL) was developed by Poole et al. (2009) to assess the impact of neuropathic pain on quality of life. The Turkish validity and reliability study was conducted by Acar et al. (2016) (Acar et al., 2016; Poole et al., 2009). In the original study, the internal consistency of the total NePIQoL was reported as 0.86, while in the validity and reliability study, it was found to be 0.99. The scale consists of five subdimensions: pain and other symptoms, relationships, daily activities, emotional impact of pain, and personal/self-care. It is a 42-item, 5-point Likert-type scale. The minimum possible score on the questionnaire is 42, while the maximum is 210. A score closer to 210 indicates a greater negative impact of neuropathic pain on quality of life. Conversely, lower scores reflect a better quality of life with less impact from neuropathic pain.

OTHER OUTCOMES:
Change in Electroneuromyography (ENMG) Parameters | Electromyography (EMG) evaluations will be conducted twice during the study
  Electroneuromyography (ENMG) assesses nerve, muscle, and motor neuron functions by converting electrical signals into interpretable data (Rabbi et al., 2019). Used in diabetic patients for over 50 years, ENMG evaluates compound muscle action potential (CMAP) and sensory nerve action potential (SNAP), mainly for diabetic neuropathy (Najafi et al., 2018). This study will assess motor conduction in the lower extremities by recording from the abductor hallucis and extensor digitorum brevis muscles via tibial and common peroneal nerve stimulation, measuring distal latency, CMAP amplitude, and conduction velocity. Sensory conduction will be tested by stimulating sural nerves 12 cm proximally from the lateral malleolus using surface (motor) and ring (sensory) electrodes (Erbas et al., 2011; Ovayolu et al., 2008; Sarılar & Gök, 2021). ENMG will be performed at room temperature with a Medelec Synergy EMG system, ensuring skin temperature >31°C, at baseline and three months later.
Visual Analog Scale (VAS) | The scale was filled in the baseline
  Clothing comfort is crucial for both manufacturers and users (Bertaux et al., 2010), with garments needing to avoid discomfort. Comfort involves various sensory aspects: visual (aesthetic), thermal (cold/heat), pain (tingling/itching), and tactile (smooth/rough, soft/hard) (Malik & Sinha, 2012; Soroka et al., 2019). Studies use objective methods (Herbaut et al., 2016; Teyeme et al., 2021) and subjective scales (Matthias et al., 2021; Mills et al., 2011). We will assess sock comfort using a Visual Analog Scale (VAS), ranging from "Very Comfortable" (10) to "Very Uncomfortable" (0). The VAS will be collected at each follow-up, with prior instructions given. Participants will consider visual, thermal, pain, and tactile properties while rating their experience.

CONTACTS AND LOCATIONS:
Locations (1):
- Erciyes Üniversitesi, Talas, Kayseri, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided